CLINICAL TRIAL: NCT02376868
Title: Topcon 3D OCT-1 Maestro Agreement and Precision Study II
Brief Title: Maestro Agreement and Precision Study II
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: MaestroAPII
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Normal Healthy Subjects With No Known Ocular Diseases; Glaucomatous Eyes; Eyes With Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal Eyes: Subjects with no known ocular diseases will be scanned with the iVue and Maestro device
  Interventions: Device: 3D OCT-1 Maestro; Device: iVue
- Glaucomatous Eyes: Subjects presenting with different stages of glaucoma will be scanned with the iVue and Maestro device
  Interventions: Device: 3D OCT-1 Maestro; Device: iVue
- Eyes with Retinal Diseases: Subjects presenting with Retinal pathological eyes will be scanned on the iVue and Maestro device
  Interventions: Device: 3D OCT-1 Maestro; Device: iVue

INTERVENTIONS:
Device: 3D OCT-1 Maestro — OCT machines used for diagnostic purposes
Device: iVue — OCT machines used for diagnostic purposes

SUMMARY:
Assess the repeatability and agreement of the Optic Disc Parameters, Retinal Nerve Fiber Layer (RNFL) Thickness, Full Retinal Thickness, and Ganglion Cell Thickness between the Maestro and iVue OCT devices.

ELIGIBILITY:
Inclusion Criteria for Normal Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes (eyes without pathology)
4. lOP <=21 mmHg bilaterally
5. BCVA 20/40 or better (each eye)
6. Both eyes must be free of eye disease

Exclusion Criteria for Normal Group

1. Subjects previously enrolled in either the Maestro AP study or the Maestro2 study
2. Subjects unable to tolerate ophthalmic imaging
3. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
4. HFA visual field (24-2 Sita Standard, white on white) result unreliable (based on manufacturer's recommendation), defined as fixation losses> 20% or false positives> 33%, or false negatives> 33%
5. Visual field defects consistent with glaucomatous optic nerve damage with at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."
6. Presence of any ocular pathology except for cataract
7. Narrow angle
8. History of leukemia, dementia or multiple sclerosis
9. Concomitant use of hydroxychloroquine and chloroquine

Inclusion Criteria for Glaucoma Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. BCVA 20/40 or better in the study eye
4. Visual field defects consistent with glaucomatous optic nerve damage based on with at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."
5. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

   1. Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles with or without disc hemorrhage;
   2. Localized abnormalities of the peripapillary retinal nerve fiber layer, especially at the inferior or superior poles; or
   3. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue

Exclusion Criteria for Glaucoma Group

1. Subjects previously enrolled in either the Maestro AP study or the Maestro2 study
2. Subjects unable to tolerate ophthalmic imaging
3. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
4. HFA visual field (24-2 Sita Standard, white on white) result unreliable, defined as fixation losses> 20% or false positives> 33%, or false negatives > 33% in the study eye
5. Presence of any ocular pathology except glaucoma in the study eye
6. History of leukemia, dementia or multiple sclerosis
7. Concomitant use of hydroxychloroquine and chloroquine

Inclusion Criteria for Retina Disease Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with retinal disease
4. lOP<= 21 mmHg in the study eye
5. BCVA 20/400 or better in the study eye
6. Diagnosis of some type of retinal pathology by investigator, may include, but not limited to: Macular Degeneration, Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Cystoid Macula Edema, and others

Exclusion Criteria for Retinal Disease Group

1. Subjects previously enrolled in either the Maestro AP study or the Maestro2 study
2. Subjects unable to tolerate ophthalmic imaging
3. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
4. Presence of glaucoma or any ocular pathology other than a Retinal pathology (e.g., cornea pathology) in the study eye
5. Narrow angle in the study eye
6. History of leukemia, dementia or multiple sclerosis
7. Concomitant use of hydroxychloroquine and chloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with no eye disease and subjects with retinal disease or glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Optic Disc Measurements (Optic Disc/Cup Size) | 1 Hour
  Reporting of the Optic Disc Size and Cup Size
Retinal Nerve Fiber Layer (RNFL) Thickness Measurements At Different Clock Hours | 1 Hour
  RNFL thickness measured at different clock hours
Full Retinal Thickness Measurements | 1 Hour
  Full Retinal Thicknesses measured in different quadrants of the scan
Ganglion Cell Thickness Measurements | 1 Hour
  Ganglion Cell Thickness measured in different quadrants of the scan

CONTACTS AND LOCATIONS:
Overall Officials: Charles Reisman, MS, Study Director — Topcon Corporation
Locations (1):
- Western University of Health Sciences, Pomona, California, United States